CLINICAL TRIAL: NCT06204419
Title: A Phase I Study to Assess the Safety, Tolerability, and Pharmacokinetics of XH-S002 After Single Ascending Doses, Multiple Ascending Doses and Evaluation of Food Effects in Healthy Volunteers
Brief Title: A Phase I Study of XH-S002 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: S-INFINITY Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-S002-101
Record Dates: First submitted 2023-12-18; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (XH-S002) (Experimental): Participants will receive XH-S002 once or twice daily on scheduled days.
  Interventions: Drug: XH-S002 （A）
- B (Placebo) (Experimental): Participants will receive matching placebo once or twice daily on scheduled days.
  Interventions: Other: Placebo（B）

INTERVENTIONS:
Drug: XH-S002 （A） — XH-S002 powder will be administered orally as per assigned treatment regimen.
  Arms: A (XH-S002)
Other: Placebo（B） — XH-S002 Placebo (matched) will be administered orally as per assigned treatment regimen.
  Arms: B (Placebo)

SUMMARY:
The purpose of the study is to assess the safety, tolerability and pharmacokinetics of XH-S002 in healthy volunteers under SAD (Single ascending dose) and MAD (Multiple ascending dose) studies. In addition, this study evaluates the food effects of XH-S002.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female healthy adult participants aged 18~45 years (inclusive);
2. Male body weight is no less than 50 kilogram (Kg), Female body weight no less than 45 Kg, and body mass index (BMI) between 16.0 and 25.0 kg/m2 (both inclusive).
3. Participants are in a good health and have no clinically significant abnormalities as per medical history, clinical symptoms, vital signs, physical examination, 12-lead ECG, chest X-ray, abdominal ultrasound and clinical laboratory tests (hematology, urinalysis, serum chemistry, coagulation function and fecal occult blood) results.
4. After having a detailed understanding on the nature, significance, possible benefits, possible inconvenience and potential risks of this clinical trial, Participants would be able to take part in this clinical trial voluntarily, communicate well with investigator, abide by protocol procedures and sign written informed consent form (ICF).
5. Participants promise no plan on fertility and donating sperm or ovum, and to take effective physical contraception (including female partner) from screening until one month after the end of the study.

Exclusion Criteria:

1. Pregnant or lactating woman, or woman with a positive pregnancy test.
2. Participants who are suspected or confirmed to be allergic to similar ingredient or any ingredients of investigational product, or participants who are allergic, or have a drug allergy history or specific allergic disorders (asthma, urticaria, eczema, etc.).
3. Participants with a medical history or a current disorder of cardiovascular, pulmonary, endocrine, renal, hepatic, gastrointestinal, dermatology, immunology, hematology, neurology and psychiatric.
4. Participants with clinically significant acute infection or concurrent severe infection (e.g., intravenous or oral antibiotics, anti-fungal or anti-viral drugs, etc.) or participant who has not recovered from infection within 2 weeks prior to screening.
5. Participants who had a history of gastroesophageal reflux, dyspepsia, chronic nausea, or chronic diarrhea (≥3 stools per day, ≥4 weeks) within 6 months before screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
To access the safety and tolerability of single ascending dosed of XH-S002 in healthy adults. | Approximately 1～2weeks
  Safety and tolerability of single dose of XH-S002 measured by number of subjects who experience AEs and potential clinically significant changes in clinical symptoms, vital signs, physical examinations, laboratory tests and ECG parameters.
To access the safety and tolerability of multiple ascending dosed of XH-S002 in healthy adults. | Approximately 1～2weeks
  Safety and tolerability of multiple dose of XH-S002 measured by number of subjects who experience AEs and potential clinically significant changes in clinical symptoms, vital signs, physical examinations, laboratory tests and ECG parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No